CLINICAL TRIAL: NCT02840773
Title: Impact of Implant-abutment Connection on Osteoimmunological Parameters in Short Implants: a Randomised Controlled Clinical Trial
Brief Title: OPG-RANKL Levels Around Short Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, PhD, DDS, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAP-03-2014
Record Dates: First submitted 2016-06-10; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Implant-abutment Connection; Microleakage; Short Implant
Keywords: RANKL; OPG; Peri-implant crevicular fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test group-baseline (Active Comparator): Press-fit implant connection was monitored at baseline
  Interventions: Other: Peri-implanter sulcus fluid sampling; Other: Probing depth; Other: Crestal bone loss; Other: Presence of bleeding on probing; Other: Plaque index levels
- Test group-12 month (Active Comparator): Press-fit implant connection was monitored at 12 month after prosthesis delivered.
  Interventions: Other: Peri-implanter sulcus fluid sampling; Other: Probing depth; Other: Crestal bone loss; Other: Presence of bleeding on probing; Other: Plaque index levels
- Control group-baseline (Active Comparator): Screw-retained connection was monitored at baseline
  Interventions: Other: Peri-implanter sulcus fluid sampling; Other: Probing depth; Other: Crestal bone loss; Other: Presence of bleeding on probing; Other: Plaque index levels
- Control group-12 month (Active Comparator): Screw-retained connection was monitored at 12 month after prosthesis delivered.
  Interventions: Other: Peri-implanter sulcus fluid sampling; Other: Probing depth; Other: Crestal bone loss; Other: Presence of bleeding on probing; Other: Plaque index levels

INTERVENTIONS:
Other: Peri-implanter sulcus fluid sampling — PISF sampling was made twice
Other: Probing depth — The change of probing depth between baseline and 12 month after prosthetic loading. Probing depth was measured with a plastic periodontal probe (mm)
Other: Crestal bone loss — Crestal bone loss was measured on digital radiographs at baseline and after 1 year of prosthetic loading with a Java program me (Image-J 3.0 NIH, Bethesda, USA)
Other: Presence of bleeding on probing — The change bleeding on probing of between baseline and 12 month after prosthetic loading. Presence of bleeding on probing were performed at four sites of implants.
Other: Plaque index levels — The change of plaque index level between baseline and 12 month after prosthetic loading. Presence of plaque index was performed at four sites of implants.

SUMMARY:
The aim of the present study was to determine the levels of sRANKL and OPG as well as their relative ratio in PICF surrounding the two different types of implant-abutment connections on short implants after a 12-month monitoring period. Additionally, their association with clinical findings and microbiological markers in plaque samples were assessed in the present study.

DETAILED DESCRIPTION:
The peri-implant crevicular fluid (PICF) contains several inflammatory mediators; the level of these mediators can provide information on the inflammatory state of the tissue, including the activation of mechanisms of bone destruction. In this context, soluble receptor activator of nuclear factor кB ligand (sRANKL) and osteoprotegerin (OPG) have been suggested as molecular determinants of bone resorption. However, currently, there are only limited studies on the molecular responses of healthy peri-implant tissues following placement of implants on function. The null hypothesis of the present study was that there are no significant differences in the levels of sRANKL and OPG in PICF or in the respective levels of six bacterial species or total bacteria levels in submucosal biofilm samples taken from TIF- and TIS-type implants. Therefore, the aim of the present study was to determine the levels of sRANKL and OPG as well as their relative ratio in PICF surrounding the two different types of implant-abutment connections on short implants after a 12-month monitoring period. Additionally, their association with clinical findings and microbiological markers in plaque samples were assessed in the present study.Thirty short implants were randomly placed in posterior maxillary edentulous sites using a split-mouth design in 15 periodontally healthy subjects. Tapered interference fit (TIF) and taper integrated screwed-in (TIS) types of implant-abutment connections were selected for investigation. PICF and submucosal biofilm samples were collected one month after surgery and repeated 12 months after prosthetic loading. Clinical parameters, including probing depth, dichotomous presence of bleeding on probing, and plaque index, were recorded and digital periapical radiographs were taken at each time point. sRANKL and OPG levels in PICF were analyzed using an enzyme-linked immunosorbent assay. Total bacterial levels, as well as levels of Fusobacterium nucleatum, Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Prevotella intermedia, and Streptococcus oralis, were analyzed in corresponding submucosal biofilm samples using quantitative real-time polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* sufficient bone height for a 6 mm implant and sufficient bone width for a minimum 5.5 mm implant without any augmentation techniques
* no history of periodontitis.

Exclusion Criteria:

* Patients with any systemic diseases
* Smokers were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peri-implanter sulcus fluid levels of RANKL | Baseline
  Peri-implanter sulcus fluid were sampled at baseline (without prosthetic loading).
Peri-implanter sulcus fluid levels of RANKL | 12 month
  Peri-implanter sulcus fluid were sampled at 1 year after prosthetic loading.
Peri-implanter sulcus fluid levels of OPG | Baseline
  Peri-implanter sulcus fluid were sampled at baseline (without prosthetic loading).
Peri-implanter sulcus fluid levels of OPG | 12 month
  Peri-implanter sulcus fluid were sampled at 1 year after prosthetic loading.

SECONDARY OUTCOMES:
Probing depth | Baseline
  The level of probing depth at baseline. Probing depth was measured with a plastic periodontal probe.
Probing depth | 12 month
  The level of probing depth at 12 month. Probing depth was measured with a plastic periodontal probe.
Bleeding on probing | Baseline
  The level of clinical parameters bleeding on probing at baseline without prosthetic loading. The presence of bleeding on probing were performed at four sites of implants after 10 sec. of probing.
Bleeding on probing | 12 month
  The level of clinical parameters bleeding on probing at 12 month after prosthetic loading. The presence of bleeding on probing were performed at four sites of implants after 10 sec. of probing.
Plaque index | Baseline
  The level of plaque index at baseline without prosthetic loading. The dichotomous presence of supra gingival plaque was recorded at four sites of implants
Plaque index | 12 month
  The level of plaque index at 12 month after prosthetic loading. The dichotomous presence of supra gingival plaque was recorded at four sites of implants
Crestal bone loss | Between baseline and 1 year after prosthetic loading
  Crestal bone loss measured by digital periapikal radiographs at same time of PISF sampling

CONTACTS AND LOCATIONS:
Overall Officials: Veli Özgen Öztürk, PhD,DDS, Principal Investigator — Ege University, School of Dentistry, Department of Periodontology
Locations (1):
- Ege University, School of Dentistry, Department of Periodontology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes